CLINICAL TRIAL: NCT02076958
Title: Implementation of Evidence-Based Cancer Early Detection in Black Churches
Acronym: Project HEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R01CA147313 (NIH)
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Information Dissemination; Evidence-Based Public Health
Keywords: Implementation; Cancer; Early detection; Faith-based; Community health advisor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional/classroom (Active Comparator): Community health advisors trained using traditional/classroom methods and provided with technical assistance/support as needed
  Interventions: Behavioral: Community Health Advisor education
- Technology (Experimental): Community health advisors trained using technology/online methods and provided minimal technical assistance/support
  Interventions: Behavioral: Community Health Advisor education

INTERVENTIONS:
Behavioral: Community Health Advisor education

SUMMARY:
The aim of the proposed project is to identify an optimal implementation strategy using a set of evidence-based interventions that aim to increase early detection of breast, prostate, and colorectal cancer among African Americans as a model. These three interventions will be packaged and interwoven into a single branded project, Project HEAL (Health through Early Awareness and Learning) which will be delivered through trained Community Health Advisors (CHA) in African-American church settings. The implementation and sustainability will be evaluated using the RE-AIM Framework. Fourteen African American churches in Prince George's County, MD will be randomized to a traditional classroom training approach or an online training approach, in which the CHA training approach and level of technical assistance is varied (in-person classroom training of CHAs + monitoring/evaluation + technical assistance and training vs. online training of CHAs + monitoring and evaluation only, respectively). By varying the training methodology and level of technical assistance, we will be able to determine what level of technical assistance leads to successful implementation and sustainability. We will also identify church organizational capacity characteristics that lead to successful implementation and sustainability. The specific aims of this research are to: (1) Package the three interventions into a single branded project (Project HEAL), develop a local cancer screening resource guide, and pilot test the materials and training. (2) Implement Project HEAL in 14 churches in Prince George's County, Maryland. We will evaluate the implementation outcomes involving treatment fidelity and identify church organizational capacity characteristics that led to successful implementation. We will compare the two implementation strategies (traditional vs. online) to determine the optimal level of technical assistance necessary for successful implementation. (3) Evaluate the sustainability of Project HEAL over a two-year period of time. We will identify church organizational capacity characteristics that led to sustainability, and compare the two implementation strategies (traditional vs. online) to determine the optimal level of technical assistance for successful sustainability.

ELIGIBILITY:
Inclusion Criteria

* Advisory Panel members: adults ages 21+
* Pastors, representing each of the 14 churches enrolled in the project: active pastor of churches enrolled in the study.
* Community Health Advisors:

  * self-identified African American
  * over 21 years of age
  * regularly attend church services
  * able to complete Project HEAL training
  * have regular access to the Internet and feel comfortable completing online training activities
  * able to recruit 30 participants for the 3-part workshop series
  * able to lead the 3-part workshop series
* Workshop participants: Self-identified African American men and women ages 40-75 for women who are able to complete self-administered paper-and-pencil surveys.

Exclusion Criteria:

* Workshop participants: Men and women who have had breast, prostate, or colorectal cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2011-03; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Adherence to program delivery protocol - Implementation of the 3-workshop series. | Up to 10 months

SECONDARY OUTCOMES:
Number of training events (workshops) | Up to 10 months
Number of CHA trainees | Baseline
Completion of CHA training | Baseline
Self-report of modifications or problems with program delivery | Up to 12 months
Number of booster CHA training sessions over two-year period | 12-month; 24-month
Change in number of survey completion from baseline to 12-month to 24-month | Baseline; 12-month; 24-month
Number of educational sessions participants attended | Up to 10 months
Change in knowledge of cancer early detection from workshop 1 to workshop 3 | Up to 10 months
Change in perceived benefits of screening | Up to 10 months
Change in perceived barriers to screening | Up to 10 months
Change in self-efficacy for screening | Up to 10 months
Change in self-report of screening from baseline to 12-month to 24-month | Baseline; 12-month; 24-month
Ratings of program | Up to 10 months
Percent of eligible congregation that enrolled in the project | Baseline
Number of participants that attended educational sessions | Up to 10 months
Enrollment of churches | Baseline
  Number agreed/total approached
Number of additional training cycles completed over two year period | 12-months; 24-months
Amount of supplemental funding church receives for additional health education over two years | 12-month; 24-month
Number of continued health education activities including cancer education over two year period | 12-month; 24-month

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Holt, PhD, Principal Investigator — University of Maryland School of Public Health
Locations (1):
- University of Maryland School of Public Health, College Park, Maryland, United States

REFERENCES:
- [Background] Holt CL, Tagai EK, Scheirer MA, Santos SL, Bowie J, Haider M, Slade JL, Wang MQ, Whitehead T. Translating evidence-based interventions for implementation: Experiences from Project HEAL in African American churches. Implement Sci. 2014 May 31;9:66. doi: 10.1186/1748-5908-9-66. PMID 24885069
- [Background] Santos SL, Tagai EK, Wang MQ, Scheirer MA, Slade JL, Holt CL. Feasibility of a web-based training system for peer community health advisors in cancer early detection among african americans. Am J Public Health. 2014 Dec;104(12):2282-9. doi: 10.2105/AJPH.2014.302237. Epub 2014 Oct 16. PMID 25320894
- [Derived] Huq MR, He X, Woodard N, Chen C, Knott CL. The role of community health advisors' cancer history in implementation and efficacy of a cancer control intervention. Health Educ Res. 2023 Jul 25;38(4):350-361. doi: 10.1093/her/cyad011. PMID 36892605
- [Derived] Holt CL, Shelton RC, Allen JD, Bowie J, Jandorf L, Zara Santos SL, Slade J. Development of tailored feedback reports on organizational capacity for health promotion in African American churches. Eval Program Plann. 2018 Oct;70:99-106. doi: 10.1016/j.evalprogplan.2018.07.002. Epub 2018 Jul 21. PMID 30041105
- [Derived] Holt CL, Tagai EK, Santos SLZ, Scheirer MA, Bowie J, Haider M, Slade J. Web-based versus in-person methods for training lay community health advisors to implement health promotion workshops: participant outcomes from a cluster-randomized trial. Transl Behav Med. 2019 Jul 16;9(4):573-582. doi: 10.1093/tbm/iby065. PMID 29955889
- [Derived] Scheirer MA, Santos SL, Tagai EK, Bowie J, Slade J, Carter R, Holt CL. Dimensions of sustainability for a health communication intervention in African American churches: a multi-methods study. Implement Sci. 2017 Mar 28;12(1):43. doi: 10.1186/s13012-017-0576-x. PMID 28351405
- [Derived] Santos SL, Tagai EK, Scheirer MA, Bowie J, Haider M, Slade J, Wang MQ, Holt CL. Adoption, reach, and implementation of a cancer education intervention in African American churches. Implement Sci. 2017 Mar 14;12(1):36. doi: 10.1186/s13012-017-0566-z. PMID 28292299
- See also: Community Health Awareness, Messages and Prevention (CHAMP) Lab — https://sph.umd.edu/research-impact/laboratories-projects-and-programs/community-health-awareness-messages-and-prevention-champ-lab